CLINICAL TRIAL: NCT06362577
Title: Post-marketing Clinical Study of Transrectal High-intensity Focused Ultrasound for Localized Prostate Cancer
Brief Title: Clinical Study of HIFU for Localized Prostate Cancer
Acronym: HIFU
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TSC202202
Record Dates: First submitted 2024-03-17; First posted 2024-04-12 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Localized Prostate Cancer
Keywords: HIFU; Localized prostate cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high-intensity focused ultrasound.: Medical records and questionnaire data will be collected from patients with localized prostate cancer treated with Sonablate® high intensity focused ultrasound (HIFU) and robot-assisted laparoscopic radical prostatectomy (RALP) at Renji Hospital, Shanghai Jiao Tong University School of Medicine from 2021 to 2023 for local ablation or resection. And make a summary analysis.Patients with localized prostate cancer treated by high-intensity focused ultrasound.This Group Have No intervention.These do not require medication。EQ-5D-5L IPSS IIEF-5 EPIC-26 ECOG Diagnostic Tests were collected at before surgery, during surgery,2 months, 6 months, 9 months, 12 months, 18 months and 24 months after patients with localized prostate cancer treated with Sonablate® high intensity focused ultrasound (HIFU) .
  Interventions: Diagnostic Test: EQ-5D-5L IPSS IIEF-5 EPIC-26 ECOG
- robot-assisted laparoscopic radical prostatectomy: Medical records and questionnaire data will be collected from patients with localized prostate cancer treated with Sonablate® high intensity focused ultrasound (HIFU) and robot-assisted laparoscopic radical prostatectomy (RALP) at Renji Hospital, Shanghai Jiao Tong University School of Medicine from 2021 to 2023 for local ablation or resection. And make a summary analysis.Patients with localized prostate cancer treated by robot-assisted laparoscopic radical prostatectomy (RALP)。This Group Have No intervention.These do not require medication。EQ-5D-5L IPSS IIEF-5 EPIC-26 ECOG Diagnostic Tests were collected at before surgery, during surgery,2 months, 6 months, 9 months, 12 months, 18 months and 24 months after patients with localized prostate cancer treated with robot-assisted laparoscopic radical prostatectomy (RALP) .
  Interventions: Diagnostic Test: EQ-5D-5L IPSS IIEF-5 EPIC-26 ECOG

INTERVENTIONS:
Diagnostic Test: EQ-5D-5L IPSS IIEF-5 EPIC-26 ECOG — Diagnostic Test were collected at before surgery, during surgery,2 months, 6 months, 9 months, 12 months, 18 months and 24 months after radical surgery

SUMMARY:
In this study, the safety and effectiveness data of Sonablate system, a transrectal high-intensity focused ultrasound therapeutic instrument, in the treatment of localized prostate cancer were collected, and the treatment conditions of patients with other methods (such as radical prostatectomy) were compared and analyzed. Observe the differences in treatment effect, survival rate, postoperative PSA, recurrence and complications.

To analyze and compare the clinical outcome, postoperative complications and tumor control of HIFU and robot-assisted laparoscopic radical prostatectomy for localized prostate cancer, and to explore the effectiveness and safety of HIFU in the treatment of localized prostate cancer, so as to provide an alternative treatment for localized prostate cancer.

DETAILED DESCRIPTION:
This observational study will collect medical history and questionnaire data before and after high intensity focused ultrasound (HIFU) or radical surgery to perform local ablation or excision of prostate cancer tissue.

This study established a cohort of relevant subjects and collected their postoperative follow-up data. The study was divided into two groups:

* Study group: Transrectal high intensity focused ultrasound (HIFU) therapy;
* Control group: robot-assisted laparoscopic radical prostatectomy (RALP). Compare and analyze the treatment status of the same period of patients treated by the study group or the control group, observe the differences in treatment effect, survival rate, postoperative PSA, recurrence and complications, and explore the effectiveness and safety of HIFU treatment for localized prostate cancer.

Electronic medical records of prostate cancer patients who received Sonablate® high intensity focused ultrasound (HIFU) and robot-assisted laparoscopic radical prostatectomy at Renji Hospital, Shanghai Jiao Tong University School of Medicine from 2021 to the end of the study were collected and analyzed. Baseline characteristics, postoperative complications and disease control rate were evaluated.In this study, patients clinically diagnosed with localized prostate cancer were classified into low - and medium-risk groups to receive local HIFU treatment or robot-assisted laparoscopic radical prostatectomy (RALP) from March 2021 to the end of the study through medical history review. Patient age, PSA value at the time of diagnosis of prostate cancer, and whether they received short-term antiandrogen therapy before treatment were collected. The changes of PSA levels in each group were dynamically observed after surgery, mp-MRI was performed under the guidance of ultrasound-guided, and the negative rate was calculated. Phoenix was defined as biochemical recurrence (PSA ≥2 ng/mL higher than the lowest point), and the patient experience (postoperative complications and quality of life) after HIFU and robot-assisted laparoscopic radical prostatic resection were compared. Write clinical evaluation report.

Patients meeting the inclusion criteria were divided into the control group [receiving robot-assisted laparoscopic radical prostatectomy (RALP)] and the study group [receiving high-intensity focused ultrasound (HIFU)]. A cohort of relevant patients was established and postoperative follow-up data were collected. The relevant outcome indicators and clinical indicators before and after treatment were compared between the two groups. To clarify the clinical value of high-intensity focused ultrasound in local treatment of localized prostate cancer, and further explore the related prognostic factors.

Subjects will be included in this study in a combination of retrospective and/or prospective manners.

ELIGIBILITY:
Inclusion Criteria:

1. Men over the age of Forty;
2. Localized prostate cancer for which transperineal template prostate biopsy or MRI targeted biopsy combined with systematic biopsy is performed;
3. Ti-T2cN0M0 disease stage; Serum psa < 20 ng/ml; Gleason score ≤7(3+4 or 4+3 or lower); Or the researcher evaluates the medium-low risk prostate cancer within T2 stage without lymph node and distant metastasis; Treatment was performed using Sonablate® transrectal high intensity focused ultrasound (HIFU) or robot-assisted laparoscopic radical prostatectomy (RALP)

Exclusion Criteria:

* Either must be "No" or the patient cannot be enrolled.

  1. The active stage accompanied by other genitourinary system infections 100 days before surgery;
  2. Men who have previously received radiation therapy;
  3. Laboratory-assessed abnormalities of renal function in the heart and liver prior to surgical treatment: ALT, AST, or serum alkaline phosphatase levels above the upper limit of 3-fold normal, coagulation disorders, other malignancies (history of other malignancies other than basal cell carcinoma or squamous skin carcinoma. Patients with a pre-operative history of malignancy that has not recurred in the last 5 years (superficial bladder cancer normally clears in 2 years) are permitted;
  4. The presence of a metal implant/stent in the urethra;
  5. Patients whose lesions were located at the anterior tip of the prostate and in front of the urethra, and other locations where the focus could not be reached or the acoustic channels were blocked by important organs;
  6. Those who were considered by the investigator to be unsuitable to participate in this clinical trial (such as patients with mental or emotional problems, patients with hearing, speaking, reading, and writing disorders, and poor compliance).

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study involved only male patients
Study Population: Medium-and low-risk prostate cancer patients without lymph node and distant metastasis within T2 period. Patients diagnosed with prostate cancer by histology or cytology; Combined with her clinical symptoms, digital rectal examination, serum prostate-specific antigen (PSA), and local imaging, it was confirmed pathologically through prostate biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative complications | before surgery, during surgery,2 months, 6 months, 9 months, 12 months, 18 months and 24 months after radical surgery
  The data were collected through medical records inquiry, consultation and questionnaire

SECONDARY OUTCOMES:
Prostate-specific antigen (PSA), PSA levels at 1 month, 3 months, and 6 months after surgery | before surgery, during surgery,1 months, 3months, 6 months after surgery,
  The PSA data was obtained by collecting postoperative PSA data at 1 month, 3 months, and 6 months.
Assessment of quality of life and sexual function spontaneously reported at 2, 6, and 12 months after surgery | before surgery, during surgery,2 months, 6 months, 9 months, 12 months, 18 months and 24 months after radical surgery
  The first indicator was erectile dysfunction, which was statistically analyzed by the three degrees of mild, moderate and severe, and evaluated by collecting the IIEF-5 scale. The score of 5-7 was severe, 8-11 was moderate, and 12-21 was mild.The second is the health description system, which describes five dimensions: mobility (mobility), Self-Care (self-care), Usual Activities (Usual Activities), Pain or discomfort (Pain/comfort), Anxiety or Depression (Anxiety/Depression), each dimension contains five levels: No difficulty, some difficulty, moderate difficulty, severe difficulty, unable to proceed/have very serious difficulty
The incidence of imaging recurrence that requires remedial or systemic treatment 12 months after surgery | before surgery, during surgery, 6 months, 12 months after surgery
  By collecting PSA data within 12 months after surgery, the incidence of imaging (mainly mp-MRI) recurrence
Failure-free survival (FFS) at 6 and 12 months postoperatively | before surgery, during surgery, 6 months, 12 months after surgery
  Failure-free survival (FFS) were collected up to 12 months after surgery.
Postoperative overall survival rate | before surgery, during surgery,2 months, 6 months, 9 months, 12 months, 18 months and 24 months after radical surgery
  Overall survival rates were collected up to 24 months after surgery.
Overall postoperative complication rate | before surgery, during surgery,2 months, 6 months, 9 months, 12 months, 18 months and 24 months after radical surgery
  Overallpostoperative complication rates were collected up to 24 months after surgery.
Number of device defects | before surgery, during surgery
  The number of perioperative device defects was counted

CONTACTS AND LOCATIONS:
Overall Officials: Xue Wei, Doctor's, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital-Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Wang yanqing, Dong bojun, Pan jiye and Zhu yinjie shared the research results with the research members of the project.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The first case is enrolled until the Study report is completed
Access Criteria: All the data in the project is available to the shared person.
URL: https://wk.test.wetrial-edc.com/